CLINICAL TRIAL: NCT01780909
Title: The Use of a Non-absorbable Marker for the Evaluation of the Gastrointestinal Transit. Evaluatie Van de Gastrointestinale Transit Aan de Hand Van de Niet-absorbeerbare Merker Paromomycine Sulfaat (Dutch Translation)
Brief Title: The Use of a Non-absorbable Marker for the Evaluation of the Gastrointestinal Transit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Bart Hens, Pharmacist, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DDD13PM
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Concentration-Time Profiles in Stomach & Intestine.
MeSH Terms: interventions — Paromomycin; Water; Domperidone; Loperamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Paromomycin Sulfate Fasted State (Experimental): Intake of Gabbroral® oral tablet formulation, which will be dissolved in a glas of 240mL water, in fasted state. Fasted state means that you have eaten nothing for 12 hours for the investigation and only have been drinking water. • After intake of the medicine at regular intervals, gastrointestinal fluids will be aspirated over 4 hours. You sit in a comfortable position in bed; eating and sleeping is not permitted (after 2 hours you have the possibility to drink some water). After 4 hours, the gastrointestinal catheters will be removed and you may eat and roam freely.
  Interventions: Drug: Paromomycin Sulfate Fasted State
- Paromomycin Sulfate Fed State (Experimental): Intake of Gabbroral® oral tablet formulation, which will be dissolved in a glas of 240mL water, in fed state. Fed state means that you have eaten nothing for 12 hours for the investigation and only have been drinking water. When you arrive at the hospital for the clinical trial, you will receive an Ensure Plus Shake, after the gastrointestinal catheters are placed. 20 minutes after the intake of the shake, you will receive the a glass of water, where Gabbroral is in dissolved. After intake of the medicine at regular intervals, gastrointestinal fluids will be aspirated over 4 hours. You sit in a comfortable position in bed; eating and sleeping is not permitted (after 2 hours you have the possibility to drink some water). After 4 hours, the gastrointestinal catheters will be removed and you may eat and roam freely.
  Interventions: Drug: Paromomycin Sulfate Fed State
- Paromomycin Sulfate w/ Domperidone (Experimental): Intake of Gabbroral® oral tablet formulation, which will be dissolved in a glas of 240mL water, in fasted state, in addition of the intake of Motilium® (API: domperidone 10 mg). Fasted state means that you have eaten nothing for 12 hours for the investigation and only have been drinking water. 20 minutes for the intake of the medicine, you will take 2 tablets of Motilium®, which stimulates the gastric emptying. After intake of the medicine at regular intervals, gastrointestinal fluids will be aspirated over 4 hours. You sit in a comfortable position in bed; eating and sleeping is not permitted (after 2 hours you have the possibility to drink some water). After 4 hours, the gastrointestinal catheters will be removed and you may eat and roam freely.
  Interventions: Drug: Paromomycin Sulfate w/ domperidone
- Paromomycin Sulfate w/ Loperamide HCl (Experimental): Intake of Gabbroral® oral tablet formulation, which will be dissolved in a glas of 240mL water, in fasted state, in addition of the intake of Imodium® (API: loperamide HCl 2 mg). Fasted state means that you have eaten nothing for 12 hours for the investigation and only have been drinking water. 20 minutes for the intake of the medicine, you will take 2 tablets of Imodium®, which has an inhibited effect on the intestine. After intake of the medicine at regular intervals, gastrointestinal fluids will be aspirated over 4 hours. You sit in a comfortable position in bed; eating and sleeping is not permitted (after 2 hours you have the possibility to drink some water). After 4 hours, the gastrointestinal catheters will be removed and you may eat and roam freely.
  Interventions: Drug: Paromomycin Sulfate w/ loperamide HCl

INTERVENTIONS:
Drug: Paromomycin Sulfate Fasted State
  Other Names: 250mg Paromomycin Sulfate (1 tablet) will be dissolved in 240mL water and will be given to the healthy volunteer
  Arms: Paromomycin Sulfate Fasted State
Drug: Paromomycin Sulfate Fed State
  Other Names: Ensure Plus shake will be given 20 minutes before intake of paromomycin sulfate.
  Arms: Paromomycin Sulfate Fed State
Drug: Paromomycin Sulfate w/ domperidone
  Other Names: Intake of 2 tablets Motilium(API domperidone) before The intake of paromomycin sulfate.
  Arms: Paromomycin Sulfate w/ Domperidone
Drug: Paromomycin Sulfate w/ loperamide HCl
  Other Names: Intake of 2 tablets Imodium (API Loperamide HCl) before The intake of paromomycin sulfate.
  Arms: Paromomycin Sulfate w/ Loperamide HCl

SUMMARY:
Aim of the study The aim of this study is to use Gabbroral® oral tablet formulation as marker for the evaluation of the gastrointestinal transit. By collecting and analyzing both gastric and intestinal fluids on different time points, the transfer dissolution can be distracted. For this study stomach fluid and intestinal fluid will be collected after oral intake of a commercially available dosing form of Paromomycin Sulfate (Gabbroral® oral tablet formulation), which is dissolved in a glas of 240mL water, in fasted or fed state. Four intake conditions will be tested on four different test days (with an intermediate period of at least 7 days).

1. intake of Gabbroral® oral tablet formulation, which will be dissolved in a glas of 240mL water, in fasted state.
2. intake of Gabbroral® oral tablet formulation in fed state.
3. Intake of 2 tablets of Motilium® (API: domperidone 10 mg) 20 minutes before the intake of Gabbroral® oral tablet formulation, which will be dissolved in a glas of 240mL water.
4. Intake of 2 tablets of Motilium® (API: loperamide HCl 2 mg) 20 minutes before the intake of Gabbroral® oral tablet formulation, which will be dissolved in a glas of 240mL water.

Conduct of the study

* The study consists of four testing days in the University Hospitals Leuven, Gasthuisberg campus.
* On each test day you come at the agreed time in fasting State to the Gastroenterology Department at UZ Leuven (Gasthuisberg, floor 0, Orange arrow). Fasted state means that you have eaten nothing for 12 hours for the investigation and only have been drinking water.
* A basic clinical anamnesis will be taken by a doctor to make sure that you are a healthy volunteer for our study. For making sure that you are HIV negative, you will undergo an HIV test. In case of a female volunteer, a pregnancy test will be taken in account to make sure you are not pregnant.
* Upon arrival at the hospital through the nose or the mouth two probes: one in the stomach and one in the gut. The position of both probes is controlled using fluoroscopy (x-ray).
* After a stabilisation period of ca. 20 min you will be asked for taking a single dose of Gabbroral® oral tablet formulation. On four different test days, with an intermediate period of at least 7 days, we will follow every one of following intake conditions:

  1. intake of Gabbroral® oral tablet formulation, which will be dissolved in a glas of 240mL water, in fasted state.
  2. intake of Gabbroral® oral tablet formulation in fed state.
  3. Intake of 2 tablets of Motilium® (API: domperidone 10 mg) 20 minutes before the intake of Gabbroral® oral tablet formulation, which will be dissolved in a glas of 240mL water.
  4. Intake of 2 tablets of Motilium® (API: loperamide HCl 2 mg) 20 minutes before the intake of Gabbroral® oral tablet formulation, which will be dissolved in a glas of 240mL water.
* After intake of the medicine at regular intervals, gastrointestinal fluids will be aspirated over 4 hours. You sit in a comfortable position in bed; eating and sleeping is not permitted (after 2 hours you have the possibility to drink some water).
* After 4 hours, the gastrointestinal catheters will be removed and you may eat and roam freely.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* age: 20-35 year

Exclusion Criteria:

* Diseases
* Acute/chronic gastrointestinal disorders
* Medication use
* Possible pregnancy
* Frequent exposure to x-ray radiation during the past year
* HIV positive

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Concentration-time profiles of the drug paromomycin sulfate in the stomach and intestine | This concentration-time profiles in the stomach and intestine will be measured for 4 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Gasthuisberg, Leuven, BE, Belgium